CLINICAL TRIAL: NCT02019069
Title: A Phase II Study of CPX-351 for Treatment of AML or Higher Risk MDS Relapsed or Refractory to Prior Therapy With Hypomethylating (HMA) Agent
Brief Title: CPX-351 in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rondeep Brar (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Rondeep Brar, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-28524; NCI-2013-01982 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEM0036 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-24 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Adult Acute Erythroid Leukemia (M6); Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia and Acute Monocytic Leukemia (M5); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Liposomal cytarabine-daunorubicin CPX-351 (Experimental): * 1st INDUCTION: Patients receive liposomal cytarabine-daunorubicin CPX-351 IV at a dose of 65 units/m2/day over 90 minutes on days 1, 3, and 5.
  * 2nd INDUCTION: Patients receive liposomal cytarabine-daunorubicin CPX-351 IV a dose of 65 units/m2/day over 90 minutes on days 1 and 3.
  * CONSOLIDATION: Beginning on day 28, patients receive liposomal cytarabine-daunorubicin CPX-351 IV a dose of 65 units/m2/day over 90 minutes on days 1 and 3.
  Interventions: Drug: liposomal cytarabine-daunorubicin CPX-351

INTERVENTIONS:
Drug: liposomal cytarabine-daunorubicin CPX-351 — Given IV
  Other Names: CPX-351

SUMMARY:
This phase 2 clinical trial studies how well CPX-351 (liposomal cytarabine-daunorubicin) works in treating patients with relapsed or refractory acute myeloid leukemia or myelodysplastic syndrome. Drugs used in chemotherapy, such as CPX-351, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Determine efficacy of CPX-351 by measuring the response rate as the sum of complete response (CR) and complete remission with incomplete count recovery (CRi) in older patients (age 60 and older) with: higher risk of myelodysplastic syndrome (MDS) who are refractory/relapsed after prior hypomethylating (HMA) therapy; subjects greater than 75 years old with higher risk MDS who are HMA relapsed/refractory who have progressed to acute myeloid leukemia (AML)); AML with refractory/relapsed disease after prior HMA therapy for AML.

SECONDARY OBJECTIVES:

1. Determine the safety of CPX-351, as the frequency of Grade 3 to 5 SAEs
2. Determine the duration of remission (DOR) following induction therapy with CPX-351.
3. Determine overall survival (OS) at 12 months.
4. Determine the early induction mortality (at 30 and 60 days) following CPX-351 following induction therapy.

OUTLINE:

Patients receive liposomal cytarabine-daunorubicin CPX-351 intravenously (IV) at a dose of 65 units/m2/day over 90 minutes on days 1, 3, and 5 of each induction cycle.

* 1st INDUCTION: Patients receive liposomal cytarabine-daunorubicin CPX-351 IV at a dose of 65 units/m2/day over 90 minutes on days 1, 3, and 5. Patients achieving a complete remission (CR) or a CR with incomplete blood count recovery (CRi) at day 14 proceed to consolidation therapy
* 2nd INDUCTION: Patients with reduced blast count not achieving a morphological leukemia free state (< 5% blasts) receive the 2nd course of induction therapy. Patients receive liposomal cytarabine-daunorubicin CPX-351 IV a dose of 65 units/m2/day over 90 minutes on days 1 and 3. Patients achieving a complete remission (CR) or a CR with incomplete blood count recovery (CRi) after the 2nd course of induction therapy proceed to consolidation therapy.
* CONSOLIDATION: Beginning on day 28, patients receive liposomal cytarabine-daunorubicin CPX-351 IV a dose of 65 units/m2/day over 90 minutes on days 1 and 3.

After completion of study treatment, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily give informed consent
* Age ≥ 60
* Pathological diagnosis of AML (by WHO criteria) or higher risk MDS (includes int-2 and high risk MDS by IPSS) along with one of the following:

  * Patients with de novo or secondary MDS with progression/refractoriness after HMA treatment who have not transformed to AML
  * Patients with MDS and prior HMA treatment for MDS who transform to AML
  * Patients with AML who are refractory/relapsed after HMA therapy for their AML are eligible
* Life expectancy > 1 month
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to adhere to the study visit schedule and other protocol requirements
* Laboratory values fulfilling the following:

  * Serum creatinine < 2.0 mg/dL
  * Serum total bilirubin ≤ 2.5 mg/dL. Note, patients with Gilbert's syndrome may have elevated bilirubin at baseline prior to diagnosis with AML or MDS. Patients with Gilbert's syndrome are included if their total bilirubin is ≤ 2 times their baseline total bilirubin.
  * Serum alanine aminotransferase or aspartate aminotransferase < 3 times ULN
* Cardiac ejection fraction ≥ 45% by echocardiography (transthoracic echocardiography) or MUGA scan
* Patients with second malignancies may be eligible at discretion of PI given acute life threatening nature of untreated AML or higher risk MDS. Patients maintained on long-term non-chemotherapy treatment, e.g., hormonal therapy, are also eligible.

Exclusion Criteria:

* Patients who have previously undergone allogeneic hematopoietic stem cell transplant will be excluded from this study
* Patients who have previously had > 368 mg/m2 cumulative dose of daunorubicin or > 368 mg/m2 daunorubicin-equivalent anthracycline therapy (for example, from prior treatment of solid tumors). See appendix for anthracycline equivalence table.
* Acute promyelocytic leukemia [t(15;17)]
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Patients who have had conventional intensive cytotoxic induction chemotherapy for treatment of specifically MDS or AML are excluded.
* Patients who have not previously been treated with HMA therapy will be excluded
* Clinical evidence of active CNS leukemia
* Patients with evidence of uncontrolled current myocardial impairment (e.g. unstable ischemic heart disease, uncontrolled arrhythmia, symptomatic valvular dysfunction not controlled on medical therapy, uncontrolled hypertensive heart disease, and uncontrolled congestive heart failure)
* Active and uncontrolled infection. Patients with an active infection receiving treatment and hemodynamically stable for 48 hours may be entered into the study
* Known active uncontrolled HIV or hepatitis C infection
* Known hypersensitivity to cytarabine, daunorubicin or liposomal products
* Known history of Wilson's disease or other copper-related disorders
* Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which in the opinion of the investigator would compromise the patient's safety or interfere with data interpretation
* Laboratory abnormalities:

  * Serum creatinine ≥ 2.0 mg/dL
  * Serum total bilirubin > 2.5 mg/dL. Note, patients with Gilbert's syndrome may have elevated bilirubin at baseline prior to diagnosis with AML or MDS. Patients with Gilbert's syndrome are excluded if their total bilirubin is > 2 times their baseline total bilirubin.
  * Serum alanine aminotransferase or aspartate aminotransferase > 3 times ULN

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rondeep Brar, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Cytarabine-daunorubicin CPX-351: * 1st INDUCTION: Patients receive liposomal cytarabine-daunorubicin CPX-351 IV at a dose of 65 units/m2/day over 90 minutes on days 1, 3, and 5.
  * 2nd INDUCTION: Patients receive liposomal cytarabine-daunorubicin CPX-351 IV a dose of 65 units/m2/day over 90 minutes on days 1 and 3.
  * CONSOLIDATION: Beginning on day 28, patients receive liposomal cytarabine-daunorubicin CPX-351 IV a dose of 65 units/m2/day over 90 minutes on days 1 and 3.
  liposomal cytarabine-daunorubicin CPX-351: Given IV
Period: Overall Study
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Age, Continuous [Median (Standard Deviation); unit: years] | 74 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: The response rate was determined as the sum of complete response calculated by adding the total complete response (CR) and complete response with incomplete count recovery (CRi). The outcome is reported as the total number without dispersion.
  * CR = less than 5% blasts; no blasts with auer rods; and no persistence of extramedullary disease, with blood count recovery to platelets ≥ 100,000/uL and ANC > 1000/uL, with transfusion independence.
  * CRi = all the parameters for CR, but platelets < 100,000/uL and/or ANC ≤ 1000/uL.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Complete Response With Incomplete Count Recovery (CRi)
Description: Complete response (CR) with incomplete count recovery (CRi) was determined as the number of participants who achieved CRi after induction therapy. The outcome is reported as the total number or participants without dispersion.
  * CR = less than 5% blasts; no blasts with auer rods; and no persistence of extramedullary disease, with blood count recovery to platelets ≥ 100,000/uL and ANC > 1000/uL, with transfusion independence.
  * CRi = all the parameters for CR, but platelets < 100,000/uL and/or ANC ≤ 1000/uL.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 1

3. Secondary Outcome: Complete Response (CR)
Description: Complete response (CR) was determined the number of participants who achieved CR by Day 42 after induction treatment. The outcome is reported as the total number of participants without dispersion.
  • CR = less than 5% blasts; no blasts with auer rods; and no persistence of extramedullary disease, with blood count recovery to platelets ≥ 100,000/uL and ANC > 1000/uL, with transfusion independence.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 2

4. Secondary Outcome: Duration of Remission (DOR) Following Induction With CPX-351
Description: Duration of remission (DOR) was assessed as the length of time from documented complete response (CR) or complete response with incomplete count recovery (CRi) until documented lost of response, relapse, or death. The outcome is reported as the median with full range.
  * CR = less than 5% blasts; no blasts with auer rods; and no persistence of extramedullary disease, with blood count recovery to platelets ≥ 100,000/uL and ANC > 1000/uL, with transfusion independence.
  * CRi = all the parameters for CR, but platelets < 100,000/uL and/or ANC ≤ 1000/uL.
  For patients remaining alive, duration of remission (DOR) is reported as the length of time from documented complete response (CR) or complete response with incomplete count recovery (CRi) until the most recent assessment.
Time Frame: Up to 1 year
Measure: Median (Full Range); unit: days
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
days | 185 [25 to 329]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed as the number of participants remaining alive 12 months, starting from date of entry into trial. The outcome is reported as the number of participants (without dispersion).
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 1

6. Secondary Outcome: Early Induction Mortality (Day 30 After 1st Induction)
Description: Early induction mortality was assessed as the number of participants who died within 30 days of completing the 1st cycle of CPX-351 (1st induction). The outcome is reported as the number of participants without dispersion.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 2

7. Secondary Outcome: Mortality at Day 60 After 1st Induction
Description: Mortality at Day 60 after 1st induction was assessed as the number of participants who died within 60 days of completing the 1st cycle of CPX-351 (1st induction). The outcome is reported as the number of participants without dispersion.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 3

8. Secondary Outcome: Participants Experiencing of Serious Adverse Events
Description: Serious adverse events per participant were assessed as serious adverse events per 21CFR§312.32 that were Grade 3 or greater, and independent of relationship to CPX-351. The outcome is reported as the number of participants that experienced any defined SAE, a number without dispersion.
Time Frame: Up to 4 weeks after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Participants | 5

9. Secondary Outcome: Serious Adverse Events
Description: Serious adverse events were assessed as serious adverse events per 21CFR§312.32 that were Grade 3 or greater, and independent of relationship to CPX-351. The outcome is reported as the total number of the defined SAEs, a number without dispersion.
Time Frame: Up to 4 weeks after completion of treatment
Population: Per protocol, the outcome only includes SAEs that are Grade 3 or greater. Adverse events that were Grade 2 or less, (eg, Grade 2 event with hospitalization) are not included.
Measure: Number; unit: Adverse events
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
Number analyzed (Participants) | 11
Adverse events | 8

ADVERSE EVENTS:
Time Frame: Up to 4 weeks after completion of treatment]
Arm/Group | Liposomal Cytarabine-daunorubicin CPX-351
All-Cause Mortality (participants affected / at risk) | 10/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Cytarabine-daunorubicin CPX-351 (N=11)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adult repiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardio-pulmonary arrest (Cardiac disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neoplasms - Other, Acute myelogenous leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Cytarabine-daunorubicin CPX-351 (N=11)
Blood and lymphatic system disorders, other - clot in cheek (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders, other - tachycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Eye disorders, other - eye itching (Eye disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain, hip (General disorders) | 1 (1)
Pain, leg (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Lung infection (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Investigations, other - fluid overload (Investigations) | 1 (1)
Hepatobiliary disorders, other - hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Anorexia (decreased food consumption) (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder, other - broken leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 3 (3)
Renal and urinary disorders, other - urinary discomfort (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (nose bleed) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders, other - chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcutaneous tissue disorders, other - multiple subcutaneous nodules (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT02019069/Prot_SAP_000.pdf